CLINICAL TRIAL: NCT03302247
Title: Depletion of Myeloid Derived Suppressor Cells to Enhance Anti PD-1 Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to accrue subjects
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-113
Record Dates: First submitted 2017-09-27; First posted 2017-10-05 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Non Small Cell Lung Cancer Stage IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Nivolumab 240mg, IV on day 1, 15 + Gemcitabine 1000mg/m2, IV on day 1, 8, 15 of 28 days cycle
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab+Gemcitabine (Experimental): Nivolumab infusion on day 1 and 15 with the addition of gencitabine on day 1, 8 and 15 of 28 day cycle
  Interventions: Biological: Nivolumab; Drug: Nivolumab+Gemcitabine

INTERVENTIONS:
Biological: Nivolumab — Monoclonal antibody against non small cell lung cancer
Drug: Nivolumab+Gemcitabine — Gemcitabine is added to the Nivolumab treatment

SUMMARY:
Metastatic non small cell lung cancer can be treated with cytotoxic chemotherapy or using recently approved immunotherapy with antibody, Nivolumab. Both the therapies have limitation due to development of tolerance or immunosuppression. This trial combines one drug from each category, immunotherapeutic Nivolumab and chemotherapeutic gemcitabine as it was reported that gemcitabine reduces immunosuppression by killing myeloid derived suppressor cells, thereby increasing the efficacy of Nivolumab.

DETAILED DESCRIPTION:
Primary Objective

• The primary objective of this proposal is to evaluate gemcitabine as a method of MDSC depletion.

Secondary Objectives

* Evaluate whether these measures result in enhanced T-cell activity and/or NK cell function and number.
* Determine the tolerability and clinical activity (including response rate and survival) of this approach.
* Correlate MDSC number with tumor PD-L1 expression

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of non-small cell lung cancer (NSCLC). Patients should have stage IV disease (AJCC 7th edition), stage IIIb disease that is not amenable to potentially curative treatment (e.g. chemoradiotherapy) or unequivocal progression in a prior irradiated field. Measurable or evaluable disease is required.
2. Fresh/ archived tumor tissue available for molecular marker testing is required for entry. A tumor block or at least 5 unstained slides must be available. As an alternative FFPE cell block that is sufficient for histologic analysis is acceptable. If a patient has had PD-L1 status previously determined with and FDA approved assay, they have met this requirement. Tissue is still requested (but not required) for further analysis
3. Age > 18 years.
4. ECOG performance status 0 or 1
5. Patients must have normal organ and marrow functions as defined below:

   White blood cells (WBC) >2,000/mcL; Platelets >100,000/mcL; Hb ≥9g/dl; Absolute neutrophil count (ANC) >1,500/mcL; Serum creatinine ≤1.5 x ULN, or

   Creatinine clearance (CrCl) ≥50 ml/min (if using Cockcroft Gault formula below):

   Female CrCl= ((140 - age in years)/(72 x serum creatinine in mg/dL)) x weight in kg x 0.85; Male CrCl= ((140 - age in years)/(72 x serum creatinine in mg/dL) x weight in kg x 1.0; AST/SGOT ≤ 3 x ULN

   Total bilirubin:

   If no known liver metastasis: total bilirubin ≤ 1.5 x institutional upper limit (ULN) (except, subjects with Gilbert Syndrome who may have total bilirubin < 3.0 mg/dl; If known metastasis: total bilirubin ≤ 5 ULN
6. Negative serum pregnancy test result in Women os Child -bearing Potential (WOCBP)
7. Prior therapies:

   * Patients without activating mutations and gene rearrangements should have received at least one prior chemotherapy regimen. Any number of prior therapies is allowed except for immunotherapy (e.g. anti PD-1, PD-L1, vaccines, CTLA-4 etc.),
   * Patients with activating mutations with known documented benefit from tyrosine kinase inhibitors should have received and demonstrated progression with that inhibitor (e.g. EGFR del 19 mutation should have been treated with gefitinib, erlotinib or afatanib etc). ALK rearrangements should have been treated with an ALK inhibitor. Patients who have progressed on these agents should be assessed, if appropriate, for resistance mutations susceptible to approved agents and treated with that agent.
   * No prior gemcitabine treatment
8. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Patients with active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
2. Patients requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
3. As there is a potential for hepatic toxicity with nivolumab, drugs with predisposition to hepatotoxicity should be used with caution in patients treated with nivolumab-containing regimen.
4. Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated without clinical or radiologic evidence of progression for 14 days prior to initiation of treatment. An MRI within 14 days of commencing therapy is required for patients with a history of brain metastases.
5. There must be no requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab.
7. Uncontrolled inter-current illness that would increase the risk of toxicity or limit compliance with study requirements. This includes but is not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situations that would limit compliance with study requirements.
8. Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the abnormal immune response that results from HIV disease.
9. Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
10. Patients who have had systemic (IV) cytotoxic chemotherapy or any other investigational agents within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. If a patient received an oral agent, treatment on study can not commence at least five half-lives of the agent have elapsed.
11. Subjects with previous malignancies (except non-melanoma skin cancers, and in situ cancers such as the following: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
12. Other active malignancy requiring concurrent intervention.
13. Subjects with any history of interstitial lung disease.
14. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab+Gemcitabine
Started | 3
Completed | 0
Not Completed | 3
Not completed — the study has closed prematurely | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab+Gemcitabine
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Macrophage Derived Suppressor Cells (MDSC) Numbers as a Result of Treatment With Gemcitabine.
Description: Immunosuppression in terms of number of circulating MDSC in the blood by comparing within each arm reduction in the number of MDSCs after each cycle of treatment
Time Frame: 2 years
Population: The study has closed prematurely. Insufficient data for analysis
Arm/Group | Nivolumab+Gemcitabine
Number analyzed (Participants) | 0

2. Secondary Outcome: Increase in T-cell Activity
Description: Evaluate if MDSC elimination by gemcitabine results in increase in T-cell activity
Time Frame: 2 years
Population: The study has closed prematurely. Data was not collected
Arm/Group | Nivolumab+Gemcitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Nivolumab+Gemcitabine
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab+Gemcitabine (N=3)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Elevated CPK (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Intractable leg pain (General disorders) | 1
Intractable right hip pain (General disorders) | 1
Intractable lower back pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab+Gemcitabine (N=3)
Anemia (Blood and lymphatic system disorders) | 3 (6)
Constipation (Gastrointestinal disorders) | 3 (8)
Nausea (Gastrointestinal disorders) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (6)
Chills (General disorders) | 2 (3)
Fever (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 3 (8)
Creatinine increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (7)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 2 (6)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Anorexia (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoantremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Renal and urinary disorders - other (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03302247/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT03302247/ICF_001.pdf